CLINICAL TRIAL: NCT06986733
Title: Study of Management Alterations Resulting From CaRi-Heart® Technology in Patients Undergoing Coronary Computed Tomography Angiography (CCTA) for the Evaluation of Coronary Artery Disease: A United States Based Multi-Centre Study
Brief Title: Study of Management Alterations Resulting From CaRi-Heart® Technology in Patients Undergoing Coronary Computed Tomography Angiography (CCTA) for the Evaluation of Coronary Artery Disease: A United States Based Multi-Centre Study (SMART-CCTA-1)
Acronym: SMART-CCTA-1
Status: Not yet recruiting | Type: Observational
Sponsor: Caristo Diagnostics Limited (Industry)
Collaborators: Arkansas Cardiology, P.A. (Network); Baptist Health, Louisville (Other); Northeast Georgia Hospital System (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMART-CCTA-1
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an assessment of the impact of CaRi-Heart® on the clinical management of patients across at least three centres in the USA. This study is an observational study, in which clinicians will be presented with a patient's CCTA scan results and relevant clinical details (such as blood test results and clinical risk factors) with the resulting clinical management recommendation recorded; they will then be presented with the results of the CaRi-Heart® analysis alongside any other relevant clinical details and any changes in clinical management recommendation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated CCTA undertaken for evaluation of coronary artery disease.

Exclusion Criteria:

* History of surgical revascularization (coronary artery bypass graft, CABG)
* CCTA undertaken for structural heart disease evaluation (e.g. transcatheter aortic valve replacement (TAVR)
* The CCTA is of poor quality or partly unanalyzable due to artifacts, such as motion-artifacts, breathing-artifacts, stack-artifacts or blooming-artifacts.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant who has had a clinically indicated analysable CCTA at the three hospital collaborators
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of CaRi-Heart® analysis on clinical decision making after CCTA in a US setting. | Two weeks from initial review to review with CaRi-Heart results
  The percentage of patients who received a change in recommended clinical management following review of their CaRi-Heart analysis.

SECONDARY OUTCOMES:
To compare patient risk stratification with CaRi-Heart® analyses against standard clinical risk assessment tools (i.e., ASCVD-PCE). | Two weeks from initial review to review with CaRi-Heart results
  The percentage of patients reclassified into a higher (or lower) risk category using the CaRi-Heart® based AI-Risk classification, when compared to standard clinical risk assessment tools (i.e., ASCVD-PCE).
Prevalence of high coronary inflammation (defined as FAI-Score in the 75th percentile) in the study population. | Two weeks from initial review to review with CaRi-Heart results
  The percentage patients who have FAI-Score above the 75th percentile.
Prevalence of high coronary inflammation in participants with a 'normal' CCTA (i.e., CADRADS 0/1 or equivalent). | Two weeks from initial review to review with CaRi-Heart results
  The percentage patients with a CADRADs score of 0-1, who have FAI-Score above the 75th percentile.
Sub-group analysis of prevalence of high coronary inflammation by clinical site and patient demographics. | Two weeks from initial review to review with CaRi-Heart results
  The percentage patients who have FAI-Score above the 75th percentile in each of the following sub-groups: geographical location, patient age, patient sex, patient ancestry.
Correlation of FAI-Score with other available diagnostic test results (e.g., hsCRP, CACS etc.). | Two weeks from initial review to review with CaRi-Heart results
  The correlation coefficient for FAI-Score versus other available diagnostic test results (e.g., hsCRP, CACS etc.).
Correlation of FAI-Score with quantitative plaque metrics (non-calcified plaque, calcified plaque, plaque burden) | Two weeks from initial review to review with CaRi-Heart results
  The correlation coefficient for FAI-Score versus the quantitative plaque metrics.

OTHER OUTCOMES:
Prevalence of MACE in population with high coronary inflammation (FAI-Score ≥ 75th percentile) vs. those without (FAI-Score < 75th centile) | Two weeks from initial review to review with CaRi-Heart results
  A comparison of the number of major adverse cardiac events (MACE) in the population with high coronary inflammation (FAI-Score ≥ 75th percentile) vs. those without (FAI-Score < 75th centile)